CLINICAL TRIAL: NCT01058239
Title: Bortezomib Plus Rituximab for EBV + Post Transplant Lymphoproliferative Disease (PTLD)
Brief Title: Bortezomib Plus Rituximab for EBV+ PTLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Jeremy Abramson, MD, Director, Lymphoma Program, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-346; X05289 (Other: Millennium)
Record Dates: First submitted 2010-01-26; First posted 2010-01-28 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Post-transplant Lymphoproliferative Disease; Solid Organ Transplant; Stem Cell Transplant (Bone Marrow Transplant); Epstein Barr Virus Infections
Keywords: bortezomib; rituximab; PTLD; EBV; transplantation
MeSH Terms: conditions — Epstein-Barr Virus Infections | interventions — Bortezomib; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab plus Bortezomib (Experimental): This is a single arm trial adding the new drug bortezomib to the standard drug rituximab
  Interventions: Drug: bortezomib; Drug: rituximab

INTERVENTIONS:
Drug: bortezomib — Given intravenously on days 1, 4, 8 and 11 of every cycle
  Other Names: Velcade
Drug: rituximab — given intravenously on days 1, 8 and 15 of Cycle 1 and on Day 1 of subsequent cycles
  Other Names: Rituxan; Mabthera

SUMMARY:
Post transplant lymphoproliferative disease (PTLD) is a type of B-cell non-Hodgkin lymphoma that occurs in patients with weakened immune systems due to immunosuppressive medications taken after organ or stem cell transplantation. This is usually related to a virus called Epstein-Barr (EPV). Rituximab is a type of drug called an "antibody" that specifically destroys both normal and cancerous B-cells, and is commonly used for PTLD. Bortezomib is a drug that has been approved by the Food and Drug Administration (FDA) to treat multiple myeloma and a B-cell non-Hodgkin lymphoma called Mantle Cell Lymphoma, and shows significant activity in lymphoma cells caused by EBV. In this research study, we hope to learn if the addition of bortezomib to rituximab treatment can increase the rate of complete remissions and cures of PTLD after organ or stem cell transplant.

DETAILED DESCRIPTION:
* Both rituximab and bortezomib will be given to participants intravenously. Each cycle of treatment will consist of 21 days. Rituximab will be given on Days 1, 8 and 15 of Cycle 1 and on Day 1 of subsequent cycles. Bortezomib will be given on Days 1, 4, 8 and 11 of every cycle. Participants will receive a maximum of 4 cycles.
* The following study procedures will be performed during each cycle throughout the study: Medical history review; Physical exam; Performance Status; Questionnaire; Blood draws and; PET/CT scans (After cycles 2, 4 and 6 only).
* After Cycle 4, if the study doctor feels the participant has had a complete response to treatment, then they will continue onto the Post-Treatment Surveillance period, which will consist of regular clinic visits over two years.
* However, if the study doctor feels the participant has had a partial response to treatment and that they may benefit from continuing, they will receive an additional two cycles of bortezomib and be given daily tablets of the antiviral drug valganciclovir to help further target EBV.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have had a prior solid organ or allogeneic stem cell transplant.
* Patients may be newly-diagnosed or relapsed after prior therapy
* Patients must have histologically confirmed CD20+ B-cell PTLD diagnosed according to WHO criteria. PTLD may be characterized as early lesions, PTLD/polymorphic, PTLD/monomorphic, or PTLD/other, all of which are eligible for this trial. B-cell PTLD must be associated with EBV as demonstrated either by detection of EBV antigens in tumor samples, or by increased EBV quantitative viral load in serum.
* Patients must have measurable disease
* 18 years of age or older
* Estimated life expectancy of > 3 months
* ECOG Performance status of 0, 1, or 2
* Adequate organ and marrow function
* Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.

Exclusion Criteria:

* Patients receiving any other study agents. Patients already on prophylactic doses of ganciclovir or valganciclovir because of a prior history of CMV infection or because of risk factors for CMV infection are eligible for the study and may continue CMV prophylaxis.
* Patients with known brain metastases or central nervous system (CNS) involvement of their lymphoma.
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to bortezomib, rituximab, ganciclovir or valgancyclovir.
* Patients with Grade 2 or greater neuropathy within 14 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women
* Individuals with a history of malignancy are ineligible except for those outlined in the protocol
* Known HIV positive individuals
* Active HBV infection may be included only if they are on appropriate anti-hepatitis B therapy and have an undetectable HBV viral load
* Patient has received other investigational drugs within 14 days before enrollment
* Prior bortezomib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Abramson, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rituximab Plus Bortezomib
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab Plus Bortezomib
Number analyzed (Participants) | 7
Age, Continuous [Median (Full Range); unit: years] | 67 [46 to 71]
Age, Customized [Count of Participants; unit: Participants]
  ≤ 50 years | 1
  51-60 years | 0
  61-70 years | 3
  71+ years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status 0: Asymptomatic (Fully active)
  1. Symptomatic but completely ambulatory (Restricted in physically strenuous activity but ambulatory and able to carry out light work)
  2. Symptomatic <50% in bed during the day (Ambulatory and capable of all self care but unable to carry out any work activities)
  3. Symptomatic, >50% in bed, but not bedbound (Capable of only limited self-care, confined to bed or chair 50% or more of waking hours)
  4. Bedbound (Completely disabled. Cannot carry on any self-care)
  5. Death
  Participants
    0 | 4
    1 | 2
    2 | 1
WHO Classification [Count of Participants; unit: Participants] — World Health Organization (WHO) disease classification.
  * PTLD: Post-transplant lymphoproliferative disease
  * DLBCL: diffuse large B-cell lymphoma.
  Participants
    PTLD/polymorphic | 2
    PTLD/monomorphic, DLBCL | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate includes both complete and partial responses assessed by PET/CT following completion of therapy. Response was evaluated using the International Working Group criteria for lymphoma response. The complete list of criteria used to evaluate response is too long to be detailed in the allotted space here, but response is defined more generally as:
  * Complete Response (CR): Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy.
  * Partial Response (PR): ≥ 50% decrease in the sum of the products of the diameters (SPD) of up to six of the largest dominant nodes or nodal masses.
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab Plus Bortezomib
Number analyzed (Participants) | 7
Participants | 3

2. Secondary Outcome: Complete Response Rate
Description: The number of participants with complete responses as assessed by PET/CT following completion of therapy. Response was evaluated using the International Working Group criteria for lymphoma response.
  Complete Response (CR): Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy.
Time Frame: 4 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab Plus Bortezomib
Number analyzed (Participants) | 7
Participants | 3

3. Secondary Outcome: Six-Month Progression Free Survival
Description: Percent of participants with progression free survival (alive without disease progression) six months after registration. Progression was evaluated using the International Working Group criteria for lymphoma response.
  > Progressive Disease (PD) or Relapsed Disease (RD):
  1. Appearance of any new lesion > 1.5 cm in any axis during or at end of therapy. Increased Radiolabeled[18F]-2-fluoro-2-deoxy-D-glucose (FDG) uptake in a previously unaffected site will be considered PD/RD only after confirmation by other modalities.
  2. ≥ 50% increase from nadir in the sum of the products of the largest diameters (SPD) of any previously involved node, or in a single involved node, or in the sizes of other lesions.
  3. ≥ 50% increase in the longest diameter of any single previously identified node > 1 cm in its short axis.
  4. PET (positron emission tomography) positive prior to therapy: post-treatment PET should be positive unless lesion is too small to be detected with current PET sys
Time Frame: six months
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab Plus Bortezomib
Number analyzed (Participants) | 7
percentage of participants | 43 [14 to 70]

4. Secondary Outcome: Overall Survival
Description: The percent of participants surviving at 6 months and 1 year.
Time Frame: 6 months, 1 year
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Rituximab Plus Bortezomib
Number analyzed (Participants) | 7
percentage of participants
  6 month | 86 [45 to 97]
  12 Month | 86 [45 to 97]

5. Secondary Outcome: Effects of Bortezomib/Rituximab on EBV Quantitative Viral Load
Description: The Mean epstein barr virus (EBV) viral load at the given time points.
Time Frame: baseline, 21, 42, 63, 84 days (end of cycles 1, 2, 3, 4)
Population: Not all participants completed four cycles of treatment. The number of participants analyzed in each row differs according to the number of participants available for analysis at each time point.
Measure: Mean (Standard Deviation); unit: Log2[(viral copies/ milliliter blood)+1]
Arm/Group | Rituximab Plus Bortezomib
Number analyzed (Participants) | 7
Log2[(viral copies/ milliliter blood)+1]
  Baseline | 13.02 (3.39)
  End of Cycle 1 (21 days): number analyzed (Participants) | 5
  End of Cycle 1 (21 days) | 10.12 (3.18)
  End of Cycle 2 (42 days): number analyzed (Participants) | 5
  End of Cycle 2 (42 days) | 9.11 (6.19)
  End of Cycle 3 (63 days): number analyzed (Participants) | 4
  End of Cycle 3 (63 days) | 8.98 (2.29)
  End of Cycle 4 (84 days): number analyzed (Participants) | 3
  End of Cycle 4 (84 days) | 7.85 (0.34)

6. Secondary Outcome: Treatment Related Toxicities
Description: The toxicities experienced by participants that were deemed to be related to the study treatment. Data is shown as the number of participants that experienced any grade toxicity that was deemed to be related to treatment. Toxicities were assessed with the use of Common Toxicology Criteria for Adverse Events (CTCAE).
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Rituximab Plus Bortezomib
Number analyzed (Participants) | 7
participants
  Febrile Neutropenia | 1
  Leukocytosis | 1
  Lymph Node Pain | 2
  Abdominal Pain | 1
  Nausea | 1
  Neutrophil Count Decreased | 2
  Platelet Count Decreased | 4
  Alkalosis | 1
  Anorexia | 1
  Peripheral Sensory Neuropathy | 2

ADVERSE EVENTS:
Time Frame: From baseline until the participant is off study, median duration of 14.9 months
Description: Adverse events were assessed with the use of regularly scheduled physical exams, laboratory tests, and patient self reports.
Arm/Group | Rituximab Plus Bortezomib
All-Cause Mortality (participants affected / at risk) | 1/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab Plus Bortezomib (N=7)
Platelet count decreased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rituximab Plus Bortezomib (N=7)
Leukocytosis (Blood and lymphatic system disorders) | 2 (3)
Cardiac arrest (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Catheter related infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (19)
Neutrophil count decreased (Investigations) | 7 (38)
Platelet count decreased (Investigations) | 7 (37)
Alkaline phosphatase increased (Investigations) | 1 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (6)
Peripheral motor neuropathy (Nervous system disorders) | 7 (37)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (37)
Urinary tract pain (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes